CLINICAL TRIAL: NCT02610608
Title: Assistance Médicale à la Procréation et Risque Thrombotique
Brief Title: Medical Assistance for the Procreation and Risk of Thrombosis.
Acronym: AMPERT
Status: Terminated | Type: Observational
Why Stopped: RECRUITMENT DIFFICULTIES
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: AMPERT (RB13.160)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Hyperstimulation Syndrome; Cardiovascular Diseases; Embolism and Thrombosis
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome; Cardiovascular Diseases; Embolism and Thrombosis | interventions — Ovulation Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One blood sample for each women particpating in the study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing ART: Observation of the incidence of venous and arterial thrombosis following ovarian stimulation
  Interventions: Other: ovarian stimulation

INTERVENTIONS:
Other: ovarian stimulation — evaluation of clincal practice regarding prevention of arterial and venous thrombosis following ovarian stimulation

SUMMARY:
This study aims at evaluating clincal practice regarding prevention of arterial and venous thrombosis following ovarian stimulation.

Secondary outcomes are : 1) to describe the incidence and risk factors of arterial and venous thrombosis in women undergoing assisted reproductive technology and 2)to identify the incidence and risk factors for ovarian hyperstimulation syndrome in these women

DETAILED DESCRIPTION:
All women undergoing an assisted reproductive tecnology in order to receive an in vitro fertilization in French centers will be included in the study. These women will be followed up until 12 months after ovarian stimulation if they get pregnant or until 3 months if the stimulation does not lead to pregnancy. Risk factors for thrombosis and ovarian hyperstimulation syndrome will be collected in each woman. At each visit, women will be asked whether arterial and/or venous thrombosis had occured.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing ovarian stimulation in order to receive in vitro fertilization

Exclusion Criteria:

* Age<18 years
* Women refusing to particpate in the study
* No health coverage
* Women under guardianship
* Women receiving therapeutic doses of anticoagulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing assisted reproductive thechnology
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2016-11-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of professional clinical practice for ovarian stimulation care | Until 12 months followin ovarian stimulation

SECONDARY OUTCOMES:
Arterial and/or venous thrombosis | until 12 months following ovarian stimulation
Risk factors for thrombosis | until 12 months following ovarian stimulation

OTHER OUTCOMES:
Incidence and risk factors for ovarian hyperstimuation syndrome | until 12 months following ovarian stimulation

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Clinique Pasteur, Brest
  - Medicentre- Clinique du Val d'Ouest, Écully
  - SELARL Gynecologia, Grenoble
  - Hôpital Saint Joseph, Marseille
  - CHU de Nice - Hôpital de l'Archet, Nice
  - AP-HP - Hôpital Bichat, Paris
  - Clinique Multualiste La sagesse, Rennes
  - Clinique Mathilde, Rouen
  - CHU de Strasbourg - CMCO, Schiltigheine